# **Statistical Analysis Plan**

**Study ID:** 213514

**Official Title of Study:** A Multicentre, Open-label, Non-comparative Phase IV Clinical Study to Evaluate the Safety and Clinical Efficacy of Augmentin Extra Strength (ES)-600 (amoxicillin/potassium clavulanate 14:1 combination) in Children with Acute Respiratory Tract Infections (ARTIs) in India

NCT Number-NCT04600752

**Approval Date of Document:** 18 Jul 2022






# STATISTICAL ANALYSIS PLAN

## 213514

A Multicentre, Open-label, Non-comparative Phase IV Clinical Study to Evaluate the Safety and Clinical Efficacy of Augmentin Extra Strength (ES)-600 (amoxicillin/potassium clavulanate 14:1 combination) in Children with Acute Respiratory Tract Infections (ARTIs) in India

AUTHOR:

VERSION NUMBER AND DATE: V1.0, 18JUL2022

\\ieedc-vnasc01\BIOSdata\GSK\BRL25000\PPD Biostatistics\Documentation\SAP Document:

Author: Version Number: V1.0 Version Date: 18JUL2022

Template No.: CS\_TP\_BS016 Revision 6 Reference: CS\_WI\_BS005




## STATISTICAL ANALYSIS PLAN SIGNATURE PAGE

Statistical Analysis Plan v1.0 (Dated 18Jul2022) for Protocol 213514/Amendment 01.

| | Name | Signature | Date (DDMMYYYY) |
|---|---|---|---|
| Author: | | Refer to eSignature | PPD |
| Position: Statistical Scientist | | | |
| Company: | IQVIA, India | | |
| Author: | D | Refer to eSignature | PPD |
| Position: | Biostatistician 1 | | |
| Company: IQVIA, India | | | |
| Author: | | Refer to eSignature | PPD |
| Position: | Biostatistician 1 | | |
| Company: | IQVIA, India | | |

Upon review of this document, the undersigned approves this version of the Statistical Analysis Plan, authorizing that the content is acceptable for the reporting of this study.

| | Name | Signature | | Date (DDMMYYYY) |
|---|---|---|---|---|
| Approved By: | PPD | | PPD | |
| Position: | Manager - Statistics | 3 | | |
| Company: | GlaxoSmithKline Pl | harmaceuticals I | .td | |
| | PPD | | PF | PD |
| Approved By: | | | | |
| Position: | Senior Manager – S | tatistics | | |
| | \BIOSdata\GSK\BRL25000\ | PPD Biostatisti | ics\Docu | mentation\SAP |
| Author: PPD | | Ver | sion Nur | nber: V1.0 |

Version Date:

Reference: CS\_WI\_BS005

18JUL2022

Effective Date: 02Dec2019

Template No.: CS\_TP\_BS016 Revision 6





Statistical Analysis Plan 

| Company: | GlaxoSmithKline Pharmaceuticals Ltd |
|----------|-------------------------------------|

Document: \\ieedc-vnasc01\BIOSdata\GSK\BRL25000\\prec{PPD} \\Biostatistics\Documentation\SAP

Author: Version Number: V1.0

Version Date: 18JUL2022

Template No.: CS\_TP\_BS016 Revision 6 Reference: CS\_WI\_BS005

Effective Date: 02Dec2019



Statistical Analysis Plan 

# MODIFICATION HISTORY

| Unique<br>Identifier<br>for this<br>Version | Date of the<br>Document<br>Version | Author | Significant Changes from<br>Previous Authorized Version |
|---|---|---|---|
| 1.0 | 18JUL2022 | PPD | Not Applicable – First Version |


Template No.: CS\_TP\_BS016 Revision 6 Reference: CS\_WI\_BS005

Effective Date: 02Dec2019




## ABBREVIATIONS

| AE | Adverse Event |
|--------|----------------------------------------------|
| ABRS | Acute bacterial rhinosinusitis |
| ALT | Alanine aminotransferase |
| AMC | Amoxicillin |
| AOM | Acute otitis media |
| ARTI | Acute Respiratory Tract Infections |
| AST | Aspartate aminotransferase |
| ATC | Anatomical Therapeutic Class |
| CABP | Community-Acquired Bacterial Pneumonia |
| CI | Confidence Interval |
| CTMS | Clinical Trial Management System |
| CVA | Clavulanic acid |
| DMC | Data Monitoring Committee |
| ECG | Electrocardiogram |
| EOT | End of Treatment |
| ENR | Enrolled Population |
| FU | Follow Up |
| ES | Extra Strength |
| ITT | Intent-To-Treat |
| MEdDRA | Medical Dictionary for Regulatory Activities |

Document: \\ieedc-vnasc01\BIOSdata\GSK\BRL25000\\prec{PPD} Biostatistics\Documentation\SAP


Template No.: CS\_TP\_BS016 Revision 6 Reference: CS\_WI\_BS005



#### Statistical Analysis Plan


| ОТ | On Therapy |
|--------|----------------------------------|
| PT | Preferred term |
| PDD | Protocol Defined Diarrhea |
| SAE | Serious Adverse Event |
| SAP | Statistical Analysis Plan |
| SOC | System Organ Class |
| TEAE | Treatment Emergent Adverse Event |
| WHO | World Health Organization |
| WHO-DD | WHO Drug Dictionary |

\\ieedc-vnasc01\BIOSdata\GSK\BRL25000\PPD Biostatistics\Documentation\SAP Document:

PPD Author: Version Number: V1.0

18JUL2022

Version Date:

Template No.: CS\_TP\_BS016 Revision 6 Reference: CS\_WI\_BS005






## TABLE OF CONTENTS

| 1. | INTRODUCTION | 10 |
|-------|------------------------------------------|--------------------|
| 2. | STUDY OBJECTIVES, ENDPOINTS AND ESTIMAND | S 10 |
| 2.1. | Primaryand Secondary Objective | 10 |
| 2.2. | Estimands | 11 |
| 3. | STUDY DESIGN | 14 |
| 3.1. | General Description | 14 |
| 3.2. | Schedule of Events | 16 |
| 3.3. | Changes to Analysis from Protocol | 16 |
| 4. | PLANNED ANALYSES | 17 |
| 4.1. | Data Monitoring Committee (DMC) | 17 |
| 4.2. | Interim Analysis | 17 |
| 4.3. | Final Analysis | 17 |
| 5. | ANALYSIS POPULATIONS | 17 |
| 5.1. | Enrolled Population [ENR] | 17 |
| 5.2. | Intent To Treat Population (ITT) | 17 |
| 6. | GENERAL CONSIDERATIONS | 18 |
| 6.1. | Reference Start Date and Study Day | 18 |
| 6.2. | Baseline | 18 |
| 6.3. | Computation of Age | 18 |
| 6.4. | Analysis Period | 19 |
| Docu | | \Documentation\SAP |
| Autho | or: PPD Versi | on Number: V1.0 |

Template No.: CS\_TP\_BS016 Revision 6

Effective Date: 02Dec2019

Copyright © 2009, 2010, 2012, 2016, 2018, 2019 IQVIA. All rights reserved. The contents of this document are confidential and proprietary to IQVIA Holdings Inc. and its subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.

Version Date:

Reference: CS\_WI\_BS005

18JUL2022





#### Statistical Analysis Plan

| 6.5. | Retests, Unscheduled Visits and Early Termination Data | 21 |
|---|---|---|
| 6.6. | Windowing Conventions | 21 |
| 6.7. | Statistical Tests | 22 |
| 6.8. | Sample Size Estimation | 22 |
| 6.9. | Software Version | 23 |
| 7. | STATISTICAL CONSIDERATIONS | 23 |
| 7.1. | Adjustments for Covariates and Factors to be Included in Analyses | 23 |
| 7.2. | Multicenter Studies | 23 |
| 7.3. | Missing data | 23 |
| 7.4. | Multiple Comparisons/ Multiplicity | 23 |
| 8.<br>9. | OUTPUT PRESENTATIONS DISPOSITION AND WITHDRAWALS | |
| 9.1. | Disposition | |
| 9.2. | Protocol Deviations | |
| 10. | DEMOGRAPHIC AND OTHER BASELINE CHARACTERIST | ICS25 |
| 11. | SURGICAL AND MEDICAL HISTORY | 26 |
| 12. | CONCOMITANT MEDICATIONS | 27 |
| 13. | STUDY MEDICATION EXPOSURE | 27 |
| 13.1. | Derivations | 28 |
| 14. | STUDY MEDICATION COMPLIANCE | 28 |
| 14.1. | Derivations | 28 |
| 15. | EFFICACY ENDPOINTS | 28 |
| 15.1. | Secondary Efficacy EndpointS | 28 |
| Docun | ment: \\ieedc-vnasc01\BIOSdata\GSK\BRL25000\PPD Biostatistics\Documer | ntation\SAD |
| Docun<br>Autho | PPD | |
| Autilo | Version Date: | 18JUL2022 |
| | version Date. | 100012022 |

Template No.: CS\_TP\_BS016 Revision 6

Effective Date: 02Dec2019

Reference: CS\_WI\_BS005



#### Statistical Analysis Plan


| 15.1.1. Analysis of Secondary Endpoint | 31 |
|---|---|
| 15.1.1.1. Clinical Response | 31 |
| 15.1.1.2. Incidence of protocol- defined diarrhoea (PDD) | 31 |
| 15.1.1.3. Patient diary endpoints | 32 |
| 16. SAFETY ENDPOINTS | 32 |
| 16.1. Adverse Events | 32 |
| 16.1.1. TEAEs: Primary Safety Endpoint | |
| 16.1.1.1. Severity | 34 |
| 16.1.1.2. Relationship to Study Medication | |
| 16.1.2. TEAEs Leading to PermanentDiscontinuation of Study Medication or Withdrawal Study | |
| 16.1.3. Serious Adverse Events | |
| 16.1.4. Adverse Events Leading to Death | |
| 16.1.5. Cardiovascular Events | 33 |
| 16.2. Deaths | 36 |
| 16.3. Laboratory Evaluations | 36 |
| 16.4. ECG Evaluations | 37 |
| 16.5. Vital Signs | 37 |
| 16.6. Other Safety Assessments | 37 |
| 17. DATA NOT SUMMARIZED OR PRESENTED | 38 |
| 18. REFERENCES | 38 |
| APPENDIX 1. PROGRAMMING CONVENTIONS FOR OUTPUTS | |
| IQVIA Output Conventions | 39 |
| Dates & Times | 39 |
| Spelling Format | 39 |
| Presentation of Treatment Groups | |
| APPENDIX 2. PARTIAL DATE CONVENTIONS | 41 |
| APPENDIX 3. SAS CODE FOR ANALYSES | |
| APPENDIX 4. MAXIMUM RECOMMENDED DOSE BY BODY WEIGHT | 43 |
| Document: \\ioadc_vnasc01\BIOSdata\GSK\BDL25000\PPD \\Biostatistics\Documentation\SAP | |
| LIGOLIMONT: MODAC-MARCOLLUICISCASTANCESCADDI DENNATORI DI MODESTINI DEL MARCOLLUICI DE LA COMPANIONI CADI | |

Document:

V1.0 Author: Version Number: Version Date: 18JUL2022

Template No.: CS\_TP\_BS016 Revision 6 Reference: CS\_WI\_BS005




## 1. Introduction

This document describes the rules and conventions to be used in the presentation and analysis of safety and clinical efficacy data for Protocol 213514. It describes the data to be summarized and analyzed, including specifics of the statistical analyses to be performed.

This statistical analysis plan (SAP) is based on protocol version 1.0 amendment 01 dated 19May2021.

# 2. STUDY OBJECTIVES, ENDPOINTS AND ESTIMANDS

#### 2.1. PRIMARYAND SECONDARY OBJECTIVE

#### Table 1

| Objectives | Endpoints |
|---|---|
| Primary | Primary |
| The primary objective of the study is to assess treatment-emergent adverse events (TEAEs) in children receiving Augmentin (ES)-600 (AMC/CVA 14:1) at 90/6.4 mg/kg/day in two divided doses, administered for 10 days in ARTIs(AOM, ABRS or CABP). | Safety will be evaluated by assessing<br>the incidences of treatment emergent<br>adverse events (TEAE). |
| Secondary | Secondary |
| The secondary objective of the study is to assess clinical efficacy and incidence of protocol defined diarrhoea (PDD) in children receiving Augmentin (ES)-600 AMC/CVA 14:1 at 90/6.4 mg/kg/day in two divided doses administered for 10 days in ARTIs (AOM, ABRS or CABP). | <ul> <li>Efficacy assessment will be based on:</li> <li>1. Early clinical response at the ontherapy visit (Day 3 to 5), defined in terms of 'success' or 'failure' to study intervention.</li> <li>2. Primary clinical response at the endof-therapy visit (Day 12 to 14), defined in terms of 'success' or</li> </ul> |

\\ieedc-vnasc01\BIOSdata\GSK\BRL25000 Document: Author:

Biostatistics\Documentation\SAP

Version Number:

V1.0

Version Date:

18JUL2022

Template No.: CS\_TP\_BS016 Revision 6 Reference: CS\_WI\_BS005




'failure' to study intervention
3. Secondary clinical response at follow-up (day 22 to 28) i.e., 'success' or 'failure'.
Incidence of protocol-defined diarrhea (PDD) in children receiving

Augmentin (ES)-600 (AMC/CVA
14:1) at 90/6.4 mg/kg/day in two divided doses administered for 10 days in ARTIs (AOM, ABRS or CABP).

## 2.2. ESTIMANDS

The primary, and secondary estimands to support regulatory decisions are described in following table:

#### Primary Estimand: -

The primary clinical question of interest is:

To assess treatment-emergent adverse events (TEAEs) in children receiving Augmentin (ES)-600 (AMC/CVA 14:1) at 90/6.4 mg/kg/day in two divided doses, administered for 10 days in ARTIS (AOM, ABRS or CABP).

The primary estimand is described by the following attributes:

Population:

Children with acute respiratory tract infections (ARTIs) in India between 6 months to 12 years of either gender

Treatment conditions:

Augmentin (ES)-600 with dose level 90/6.4 mg/kg/day twice daily (12 hourly) for 10 days.

Variables/Endpoints:

Treatment emergent adverse events (TEAEs), Serious treatment emergent adverse events (TESAEs).

Summary measure:

Document: \\ieedc-vnasc01\BIOSdata\GSK\BRL25000 \bigcirc \text{PPD} \\Biostatistics\Documentation\SAP \\
Author: \text{Version Number: V1.0} \\

Template No.: CS\_TP\_BS016 Revision 6 Reference: CS\_WI\_BS005




Counts and percentages for incidence of TEAEs and TESAEs, 95% CI for subjects who have at least one or Any TEAE.

Intercurrent events (ICEs):

Discontinuation of study treatment due to any reason – While-on-treatment strategy for TEAEs and TESAEs.

#### Rationale for Estimand:

The rationale of the while-on-treatment strategy is to estimate the occurrence of TEAEs and TESAEs when subjects have taken the dose/treatment condition.

Treatment Policy will be used for post-treatment AEs, Pre- and Post- treatment SAEs.

The reasoning of treatment policy (as collected) is to estimate the occurrence of post-treatment AEs, and pre- and post-treatment SAEs until subjects are on study will be collected and reported.

No intercurrent event is defined for other safety endpoints. The data will be analyzed as collected.

#### Secondary Estimands :-

The secondary clinical questions of interest are:

To assess Early and Primary responses in children receiving Augmentin (ES)-600 (AMC/CVA 14:1) at 90/6.4 mg/kg/day in two divided doses administered for 10 days in ARTIs (AOM, ABRS or CABP).

The secondary estimands are described by the following attributes:

- Early clinical response at on-therapy [(OT) (Day 3 to 5)]
- Population:

Children with acute respiratory tract infections (ARTIs) in India between 6 months to 12 years of either gender.

Treatment conditions:

Augmentin (ES)-600 with dose level 90/6.4 mg/kg/day twice daily (12 hourly) for 10 days.

Variable/Endpoint:

Proportion of successful early clinical response at on-therapy (OT) visit.

Summary measure:

Counts and percentages for early clinical response at on-therapy (OT) visit with corresponding 95%CI.

Intercurrent events (ICEs):

\\ieedc-vnasc01\BIOSdata\GSK\BRL25000\PPD Biostatistics\Documentation\SAP Document: PPD Author: Version Number: V1.0 Version Date: 18JUL2022 Template No.: CS\_TP\_BS016 Revision 6 Reference: CS\_WI\_BS005




 Discontinuation of study treatment due to AE, discontinuation of study treatment due to lack of efficacy and use of rescue medication - Composite strategy

If subject discontinue due to above mentioned ICEs, then early response for that subject will be imputed as a failure.

Discontinuation of study treatment due to any other reason – Treatment Policy

#### Rationale for estimand:

Discontinuation of study treatment due to AE, discontinuation of study treatment due to lack of efficacy and use of rescue medication will affect the early clinical response thus the early clinical response will be counted as failure under composite strategy.

The reasoning of treatment policy is to estimate the early clinical response until subjects are on study will be collected and reported (regardless of the intercurrent event occurring).

- Primary clinical response at end of therapy [EOT (Day 12 to 14)]
- Population:

Children with acute respiratory tract infections (ARTIs) in India between 6 months to 12 years of either gender.

Treatment conditions:

Augmentin (ES)-600 with dose level 90/6.4 mg/kg/day twice daily (12 hourly) for 10 days.

Variable/Endpoint:

Proportion of successful primary clinical response at end of therapy (EOT) visit.

Summary measure:

Counts and percentages for primary clinical response at end of therapy (EOT) visit with corresponding 95%CI.

- Intercurrent events (ICEs):
- Lack of compliance (<80%) Principal stratum</li>

Only those subjects who have at least  $(\geq)$  80% compliance would be considered in the calculation for proportion of primary clinical response

 Discontinuation of study treatment due to AE, discontinuation of study treatment due to lack of efficacy and use of rescue medication - Composite strategy

Document: \\ieedc-vnasc01\BIOSdata\GSK\BRL25000\\PPD \\Biostatistics\Documentation\SAP \\
Author: \quad \text{Version Number:} \quad \text{V1.0} \\
\quad \text{Version Date:} \quad \text{18JUL2022}

Template No.: CS\_TP\_BS016 Revision 6 Reference: CS\_WI\_BS005

Effective Date: 02Dec2019




for that subject will be imputed as a failure.

If subject discontinue due to above mentioned three ICEs, then primary clinical response

- Discontinuation of study treatment due to any other reason - Treatment Policy

#### Rationale for estimand:

Lack of compliance (<80%) will impact on primary clinical response therefore subjects who have at least (≥) 80% would be considered for primary clinical response under principal stratum strategy.

Discontinuation of study treatment due to AE, discontinuation of study treatment due to lack of efficacy and use of rescue medication will affect the primary clinical response thus the primary clinical response will be counted as failure under composite strategy.

The reasoning of treatment policy is to estimate the primary clinical response until subjects are on study will be collected and reported (regardless of the intercurrent event occurring).

No intercurrent event is defined for secondary clinical response endpoint as no events are expected to occur during the follow-up period. The data will be analyzed as collected. No intercurrent event is defined for Protocol-defined diarrhoea (PDD) endpoint. The data will be analyzed as collected.

# 3. STUDY DESIGN

# 3.1. GENERAL DESCRIPTION

This study is an open label, multi-centre, non-comparative study. Subjects will be children aged between 6 months to 12 years, presenting with ARTIs including AOM, ABRS and CABP.

At Preliminary Visit (Day 0) after signing the inform consent form by the parent/guardian and assent form by children between 7 to 12 years of age, a series of screening evaluations will be performed in order to determine whether prospective study participant meets the inclusion criteria. Enrolled and screen passed subjects will receive Augmentin (ES)-600 at 90/6.4 mg/kg/day administered in two divided doses, every 12 hours with food for 10 days.

The incidence of protocol-defined diarrhoea will be determined from information collected from the Patient Diary cards, which will be appropriately translated for all languages required based on sites participating in the trial.

Template No.: CS\_TP\_BS016 Revision 6 Reference: CS\_WI\_BS005

Effective Date: 02Dec2019




coordinated effort.



After a minimum of two treatment days (four doses) of study intervention has been taken, an 'on-therapy' (OT) visit will be scheduled between Day 3 and 5. During this visit, the investigator/study coordinator shall assess safety (primary endpoint) and 'early clinical response' (secondary endpoint). Safety parameter includes treatment emergent adverse events (TEAEs) for primary study objective. Additionally, clinical status, study intervention compliance, completion of Patient Diary cards, and concomitant medications use will also be assessed. The Investigator will assess safety parameters and clinical status whereas study coordinator will check other parameters with

Subjects with clinical 'failure' or having PDD or severe AE or SAE at OT visit (Day 3 to 5), will be withdrawn from the study intervention (as per Investigator discretion) and treated appropriately. In such case, the OT visit will be considered as End of Therapy (EOT), and all evaluations that are planned at scheduled EOT (Day 12 to 14) will be completed in this visit. However, these Subjects will return at FU visit (Day 22 to 28) for safety assessment.

Subjects with clinical 'failure' or having PDD or severe AE or SAE after OT visit (Day 3 to 5) but prior to EOT, will be scheduled to return to the site for an interim evaluation, within 24 hours of notification to the Investigator. Subjects will then be withdrawn from the study intervention (as per Investigator discretion) and treated appropriately. In such case, the interim visit will be considered as EOT visit, and all evaluations that are planned at scheduled EOT (Day 12 to 14) will be completed in this visit. However, these Subjects will return at FU visit (Day 22 to 28) for safety assessment.

The Subjects continuing in the study will return for the scheduled 'end of therapy' (EOT) evaluation between Day 12 and 14. The Investigator will enquire the participant or parent/legal guardian about development of AEs and use of concomitant medication(s).

The Investigator will perform safety (primary endpoint) and primary clinical response (secondary endpoint) evaluation. Patient Diary cards and unused medication will be returned at this visit.

Subjects who experience recurrence of signs/symptoms *after* EOT visit (Day 12 to 14), but prior to scheduled FU visit (Day 22 to 28) will be required to visit the study site twice post EOT - once for the interim visit at the time of any recurrence (Day 15 to 21) and for the scheduled FU visit (Day 22 to 28). At the interim visit, all the evaluations

which are to be performed at scheduled FU visit will be conducted. However, in such cases, all evaluations except secondary clinical response will be repeated at scheduled FU visit (Day 22 to 28). All Subjects experiencing recurrence post EOT will be treated according to the Investigator's discretion

Template No.: CS\_TP\_BS016 Revision 6 Reference: CS\_WI\_BS005




All Subjects, including withdrawals or clinical 'failures' at EOT or had disease recurrence after EOT, will return for scheduled FU visit on Day 22 to 28. This visit is required for safety assessment and administration of additional medication, if warranted.

The Subjects continuing in the study will return for the scheduled 'follow-up' (FU) visit between Day 22 and 28. The visit be considered as 'end of study' visit, where the Investigator will perform final safety (primary endpoint) and secondary clinical response (secondary endpoint) evaluation (except for recurrence) during the visit.

In general, FU visit at Day 22 to 28 includes both safety and efficacy assessment for Subjects who were clinical 'success' at EOT, but only safety assessment for the Subjects who were clinical 'failures' at EOT or had disease recurrence after EOT. These Subjects are, by definition, clinical failures at follow-up visit.

Table 2: Study Flow Chart



#### 3.2. SCHEDULE OF EVENTS

Schedule of events can be found in Section 1.3 of the protocol.

#### 3.3. CHANGES TO ANALYSIS FROM PROTOCOL

There is no change in analysis from protocol.

\\ieedc-vnasc01\BIOSdata\GSK\BRL25000\PPD Biostatistics\Documentation\SAP Document: Author: Version Number: V1.0 Version Date: 18JUL2022 Template No.: CS\_TP\_BS016 Revision 6 Reference: CS\_WI\_BS005

Effective Date: 02Dec2019




# 4. PLANNED ANALYSES

#### 4.1. DATA MONITORING COMMITTEE (DMC)

There will be no DMC for this study.

#### 4.2. INTERIM ANALYSIS

There will be no Interim analysis for this study.

#### 4.3. FINAL ANALYSIS

All analyses identified in this SAP will be performed by IQVIA Biostatistics following Sponsor Authorization of this Statistical Analysis Plan and Database Lock.

## 5. ANALYSIS POPULATIONS

The following analysis population will be defined for this study:

#### 5.1. ENROLLED POPULATION [ENR]

The all subjects enrolled (ENR) population will contain all subjects who provide informed consent for this study.

This analysis population will be used to summarize subject disposition (screen failures and reason for screen failure).

#### 5.2. INTENT TO TREAT POPULATION (ITT)

All Subjects who are enrolled and receive at least 1 administration of the investigational product (Augmentin [ES]-600) will be included in the intent-to treat population. The ITT population will be used for all safety and efficacy analyses.

\\ieedc-vnasc01\BIOSdata\GSK\BRL25000 PPD Biostatistics\Documentation\SAP Document: Author: Version Number: V1.0 Version Date: 18JUL2022

Template No.: CS\_TP\_BS016 Revision 6 Reference: CS\_WI\_BS005




## 6. GENERAL CONSIDERATIONS

#### REFERENCE START DATE AND STUDY DAY 6.1.

Study Day will be calculated from the reference start date and will be used to show start/stop day of assessments and events.

Reference start date is defined as the day of the first dose of study medication, (Day 1 is the day of the first dose of study medication) and will appear in every listing where an assessment date or event date appears.

If the date of the event is on or after the reference date, then:

Study Day = (date of event - reference date) + 1.

If the date of the event is prior to the reference date then:

Study Day = (date of event - reference date).

In the situation where the event date is partial or missing, Study Day, and any corresponding durations will appear partial or missing in the listings.

#### 6.2. BASELINE

The baseline values (non-missing) for each parameter will be the last available assessment result prior to the first dose of study administration. In case first dose can be given on Day 0 (after laboratory test result availability), the same will be considered as Day 1.

- Change from Baseline = Post-Dose Visit Value Baseline
- Percentage Change from Baseline = 100 x [(Post-Dose Visit Value Baseline) / Baseline

#### 6.3. COMPUTATION OF AGE

Each subject's age will be calculated based on their date of birth relative to the date of the preliminary visit. Where only a subject's year of birth is collected, their date of birth will be imputed with 30th June (30 Jun YYYY).

\\ieedc-vnasc01\BIOSdata\GSK\BRL25000\PPD Biostatistics\Documentation\SAP Document: PPD Author: Version Number: V1.0 Version Date: 18JUL2022 Reference: CS\_WI\_BS005 Template No.: CS\_TP\_BS016 Revision 6



 Statistical Analysis Plan

#### 6.4. ANALYSIS PERIOD

The following analysis periods are defined for this study:

- Pre-treatment period = Date of Preliminary Visit (Day 0) to Date of first dose 1
- On-treatment period = Date of first dose to Date of last dose inclusive +1
- Post-treatment period = End of last dose +1 days to End of study date

#### Treatment Period for Adverse Events:

## Pre-Treatment AE's:

An AE will be said to be pre-treatment AE if AE Start Date < Study Treatment Start Date

#### Treatment Emergent Adverse Event:

An AE will be defined as Treatment emergent adverse event (TEAE) if the AE start date is on or after treatment start date & on or before treatment stop date +1

Study Treatment Start Date  $\leq$  AE Start Date  $\leq$  Study Treatment Stop Date +1

If the last dose of study drug is missing and the AE start date is on or after the first dose of study drug, then the AE will be considered as TEAE

If the AE start date is missing or partial then the AE will be considered TEAE unless there is evidence to the contrary (e.g. month/year of onset date is present and is earlier than the month/year of first dose of study medication).

#### Post Treatment AE's:

An AE will be defined as post treatment AE if the AE start date is after the treatment stop date

AE Start Date > Study Treatment Stop Date +1

#### Duration of adverse event:

(AE resolution date – AE onset or start date ) +1

#### <u>Treatment Emergent Adverse Event (TEAE):</u>

\\ieedc-vnasc01\BIOSdata\GSK\BRL25000\PPD Biostatistics\Documentation\SAP Document: Author: Version Number: V1.0 Version Date: 18JUL2022

Template No.: CS\_TP\_BS016 Revision 6 Reference: CS\_WI\_BS005

Effective Date: 02Dec2019



During treatment Period + lag time of 1day.

Onset Time Since 1st Dose (Days):

If Treatment Start Date > AE Start Date:

Onset Time = AE Onset Date - Treatment Start Date

If Treatment Start Date < AE Onset Date:

Onset Time = AE Onset Date - Treatment Start Date +1

#### Study/Treatment Period for Concomitant medication

#### Pre-Treatment Period:

If con-med start date < date of Visit 1 (or con-med date is missing)

#### On-Treatment Period:

If Con-med start date < study treatment start date (or Con-med start date is missing) and con-med stop date ≥ study treatment start date (or Con-med start date is missing), or

If study treatment start date  $\leq$  Con-med start date  $\leq$  study treatment stop date+1.

If the study treatment stop date is missing and the con-med start date is on or after the study treatment start date, then the con-med will be on-treatment.

If the con-med start or stop date is missing or partial, then the con-med will be considered ontreatment unless there is evidence to the contrary (e.g. month/year of con-med stop date is present and is before the month/year of study treatment start date).

#### Post -Treatment Period:

If con-med stop date is after the treatment stop date+1

Con-med Stop Date > Study Treatment Stop Date+1

#### Definition of on-set for an Event:

Con-med duration (Days):

Con-med Stop Date - Con-med Start Date + 1

Time Since 1st Dose (Days):

If Treatment Start Date > Con-med Start Date:

Time = Con-med Start Date - Treatment Start Date

Document: \\ieedc-vnasc01\BIOSdata\GSK\BRL25000\\ PPD \\ Version Number: V1.0 \\ Version Date: 18JUL2022

Template No.: CS\_TP\_BS016 Revision 6 Reference: CS\_WI\_BS005

Effective Date: 02Dec2019

Copyright © 2009, 2010, 2012, 2016, 2018, 2019 IQVIA. All rights reserved. The contents of this document are confidential and proprietary to IQVIA Holdings Inc. and its subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.




 Statistical Analysis Plan

If Treatment Start Date ≤ Con-med Start Date:

Time = Con-med Start Date - Treatment Start Date +1

If Treatment Start Date or start date of Con-med is missing Time = missing.

# 6.5. RETESTS, UNSCHEDULED VISITS AND EARLY TERMINATION DATA

For by-visit summaries, refer Section 6.6 (visit windows).

Listings will include scheduled, unscheduled, retest and early discontinuation data.

#### 6.6. WINDOWING CONVENTIONS

The following visit window will be used for efficacy as well as safety assessment.

| Visit | Target<br>Days | Visit Window |
|---|---|---|
| Baseline | 0 | Prior to first dose of study medication |
| Visit 1 | 1 | #1 |
| On-therapy visit or OT visit | 3 | 2-5 |
| End of therapy visit or EOT visit | 12 | 6-14 |
| Interim visit recurrence | 18 | 15-21 |
| Follow-up visit | 25 | ≥22 |

<sup>#</sup> Visit 1 will be considered as baseline for patient diary card assessments if subject does not have patient diary data prior to Visit 1.

If there is more than one record for a given parameter within a specific visit window, then the nonmissing record closest to the target day will be summarized. If there are multiple records on the same day for a parameter, then the average value will be considered for continuous parameters, and the worst value will be considered for the categorical parameters.

Document: \\ieedc-vnasc01\BIOSdata\GSK\BRL25000\PPD Biostatistics\Documentation\SAP Author: Version Number: V1.0 Version Date: 18JUL2022

Template No.: CS\_TP\_BS016 Revision 6 Reference: CS\_WI\_BS005

<sup>\*</sup> Interim visit (< 24 hrs of notification) is required only if subject having clinical failure or PDD or server AE of SAE after OT visit prior to EOT visit. In this case all assessment of interim visit will be mapped to EOT visit as scheduled.




Study treatment discontinuation and unscheduled visit will also be considered for deriving the visit window for parameters.

#### 6.7. STATISTICAL TESTS

The default significant level will be 5%. All confidence intervals will be computed at 95% and all tests will be two-sided, unless otherwise specified in the description of the analyses.

#### 6.8. SAMPLE SIZE ESTIMATION

A total of 310 subjects will be enrolled and dosed. These 310 participants will be enrolled for each indication based on the respective prevalence as mentioned in the table below. These prevalence values are based on all ARTIs in India.

| Study | Indication | Prevalence % |
|----------------------|------------|-------------------|
| Kumari et al (2016) | AOM | 17.6 |
| Acharya et al (2003) | CAP | 8.6 (0.5% severe) |
| Shahid et al (2012) | ABRS | 14 |

The approximate ratio of samples in each indication will be 18:9:14 (AOM: CABP:ABRS). Based on this ratio, at least 136 subjects with AOM, 68 with CABP and 106 with ABRS will be enrolled for the study.

If the proportion of participants reporting at least one TEAE is 37.9% (as observed in Young et al, 2003), and assuming a sample size of 310 participants, it is estimated that the width of the 95% confidence interval would be within +/- 5.43% of the sample proportion (ie, [32.5%, 43.3%]), which equates to the lower and upper bounds of the 95% confidence interval lying within approximately 14% of the estimated proportion.

The sensitivity of the precision is calculated with respect to 5 different proportions estimated as presented below:

| Proportion estimate | Sample size | Precision | 95% CI |
|---------------------|-------------|-----------|----------------|
| 30% | 310 | 5.10% | (24.9%, 35.1%) |
| 35% | 310 | 5.31% | (29.7%, 40.3%) |
| 37.9% | 310 | 5.43% | (32.5%, 43.3%) |

Document: \\ieedc-vnasc01\BIOSdata\GSK\BRL25000\\preced{PPD} Biostatistics\Documentation\SAP

Version Number: V1.0


Template No.: CS\_TP\_BS016 Revision 6 Reference: CS\_WI\_BS005

Effective Date: 02Dec2019

Statistical Analysis Plan


| 40% | 310 | 5.45% | (34.5%, 45.5%) |
|-----|-----|-------|----------------|
| 45% | 310 | 5.54% | (39.5%, 50.5%) |
| 50% | 310 | 5.57% | (44.4%, 55.6%) |

#### 6.9. SOFTWARE VERSION

All analyses will be conducted using SAS version 9.4 or higher.

# 7. STATISTICAL CONSIDERATIONS

Continuous data will be summarized using the number of subjects (n), arithmetic mean (mean), standard deviation (SD), median, minimum value (min), and maximum value (max) values unless otherwise specified. Categorical variables will be summarized using the frequency counts (n) and percentages (%) for each possible value. Data from unscheduled visits will be included in the by-subject listings.

# 7.1. ADJUSTMENTS FOR COVARIATES AND FACTORS TO BE INCLUDED IN ANALYSES

This section is not applicable for this study.

## 7.2. MULTICENTER STUDIES

This study will be conducted by multiple investigators at multiple centers.

#### 7.3. MISSING DATA

Missing data will not be imputed in this study.

#### 7.4. MULTIPLE COMPARISONS/ MULTIPLICITY

There is no multiplicity adjustment planned for this study.

Document: \\ieedc-vnasc01\BIOSdata\GSK\BRL25000\\ PPD \\ Version Number: \text{V1.0} \\ Version Date: \text{18JUL2022}

Template No.: CS\_TP\_BS016 Revision 6 Reference: CS\_WI\_BS005




## 8. OUTPUT PRESENTATIONS

APPENDIX 1 shows conventions for presentation of data in outputs.

The templates provided with this SAP describe the presentations for this study and therefore the format and content of the summary tables, figures, and listings to be provided by IQVIA Biostatistics

## 9. DISPOSITION AND WITHDRAWALS

All subjects who provide informed consent will be accounted for in this study.

#### 9.1. DISPOSITION

Subject disposition will be summarized based on the ITT population by overall and indication. The following summaries will be included in the disposition table:

- Total number of subjects enrolled in the ITT population
- Number of subjects who completed the study treatment
- Number of subjects who completed the study
- Number and percentage of subjects who discontinued from the study
- Number and percentage of subjects who pre-maturely discontinued the study treatment as well as from the study along with reason for discontinuation.

Percentages will be based on the number of subjects in the ITT population.

A summary of reasons for screen failure and the number of subjects included in ITT population by overall and indication will be presented separately based on the enrolled population. The percentages will be based on the number of subjects in the All Enrolled analysis population.

In addition, summary of visits impacted by COVID-19 pandemic will be generated based on the ITT population by overall and indication.

Subject listings of reasons for study withdrawal, treatment discontinuation and reasons for screen failures for each indication will be provided using ITT and enrolled population respectively.

\\ieedc-vnasc01\BIOSdata\GSK\BRL25000\PPD Biostatistics\Documentation\SAP Document: Author: Version Number: V1.0 Version Date: 18JUL2022

Template No.: CS\_TP\_BS016 Revision 6 Reference: CS\_WI\_BS005






#### 9.2. PROTOCOL DEVIATIONS

Protocol deviations are the deviations from the procedure outlined in the protocol. All the important protocol deviations (PDs) will be summarized using ITT population as obtained from Clinical Trial Management System (CTMS) logs. PDs will be identified and discussed with the Investigator/Sponsor in PD review discussion and to finalize analysis set assignment.

Summary of important protocol deviations related to COVID-19 pandemic will also be provided by overall and indication using ITT population.

A subject listing of important protocol deviations identified by the study team will be presented each indication.

#### 10. DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

The following demographic data and other baseline characteristics will be presented for the ITT population by overall and indication:

- Derived Age (years)
- Age in categories ( $\leq$  6 months,  $\geq$  6 months and  $\leq$  2 years,  $\geq$  2 years and  $\leq$  5 years, ≥5 years and < 8 years, ≥8 years)
- Sex
- Race
- Ethnicity
- Weight (kg)
- Weight in categories ( $\leq 12 \text{kg}$ , > 12 kg and  $\leq 23 \text{ kg}$ , > 23 kg and  $\leq 40 \text{ kg}$ , > 40 kg)
- Height (cm)

Baseline characteristics will include vital signs parameters, bowel movements, and radiological assessments (X-Ray of chest and nasal/paranasal sinus), as performed at the time of preliminary visit.

Continuous demographic and baseline characteristics data will be summarized using descriptive statistics. For categorical data, counts and percentage of subjects in each category will be provided.

Subjects listing of demographic characteristics by indication will be provided for ITT population.

\\ieedc-vnasc01\BIOSdata\GSK\BRL25000 PPD Biostatistics\Documentation\SAP Document: PPD Author: Version Number: V1.0 Version Date: 18JUL2022

Template No.: CS\_TP\_BS016 Revision 6 Reference: CS\_WI\_BS005




## Baseline Signs and Symptoms:

The following summaries will be generated for baseline signs and symptoms with counts and percentages -

- Baseline signs and symptoms by indication using ITT population
- Baseline signs and symptoms by severity and indication using ITT population

By-subjects listing of baseline sign and symptoms by indication will be generated.

#### Baseline Bowel Habits:

The following summaries will be generated for baseline bowel habits-

- Descriptive statistics (n, mean, standard deviation, median, minimum, and maximum) on frequency of bowel movements at baseline by indication overall and indication using ITT population
- Summary (counts and percentages) and Descriptive statistics (n, mean, standard deviation, median, minimum, and maximum) on consistency of bowel movements at baseline by indication overall and indication using ITT population

Subject listing of radiographic evaluation by indication will be produced.

#### 11. SURGICAL AND MEDICAL HISTORY

Medical History conditions are defined as those conditions which stop prior to or at preliminary visit. Medical history will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) version 24.1 and will be summarized by system organ class (SOC) and Preferred Term (PT) with counts and percentages based on the intent to treat analysis population. A subject having more than one medical condition/disease within the same SOC/PT will be counted only once for that SOC or PT

Medical history will be sorted by descending order of system organ class (SOC) and total frequency of preferred term (PT) within each system organ class (SOC).

Past and current medical conditions will also be summarized with counts and percentages using ITT population by overall and indication.

Document: \\ieedc-vnasc01\BIOSdata\GSK\BRL25000\\preced{PPD} Biostatistics\Documentation\SAP


Template No.: CS\_TP\_BS016 Revision 6 Reference: CS\_WI\_BS005






#### CONCOMITANT MEDICATIONS 12.

Pre-treatment medication is defined as any medication that started and stopped prior to the first dose of study drug.

Concomitant medication is defined as any medication which started before the first dose of study drug AND was ongoing at the time of the first dose of study drug, or started on or after the date of first dose of study drug.

Medications with partially or completely missing start and/or stop dates will be handled as described in Section 6.4.

All medications will be coded using the World Health Organization (WHO) Drug Global dictionary version B3 September 2021.

Concomitant medications will be summarized using anatomical therapeutic class (ATC) level1 and ingredient by overall and indication for pre-, on and post- treatment based on the ITT analysis population. A subject having more than one medication within the same ATC Level 1 or ingredient will be counted only once for that ATC Level 1 or ingredient. Subjects listings will be provided for concomitant medications.

Concomitant medications will be sorted in descending order of total incidence across Augmentin ES treatment group for the ATC level 1 and in descending order of total incidence for the ingredient within each ATC level 1 class.

#### 13. STUDY MEDICATION EXPOSURE

Exposure to study medication in days will be presented for the ITT population.

The total exposure to Augmentin Extra Strength (ES)-600 (amoxicillin/potassium clavulanate 14:1 combination) is calculated based on derivation as mentioned in section 13.1. Subjects who entered treatment period but did not report any treatment dates will be categorized as having zero days of exposure.

Descriptive statistics summary on extent-of-exposure by overall and indication will be presented for study medication exposure using ITT population.

Subject listing of exposure for study medication by indication will also be generated.

\\ieedc-vnasc01\BIOSdata\GSK\BRL25000 PPD Biostatistics\Documentation\SAP Document: PPD Author: Version Number: V1.0 Version Date: 18JUL2022 Template No.: CS\_TP\_BS016 Revision 6 Reference: CS\_WI\_BS005


## 13.1. DERIVATIONS

Duration of exposure days = (date of last study drug administration – date of first study drug administration) + 1.

## 14. STUDY MEDICATION COMPLIANCE

Subject compliance will be assessed by measuring the number of doses per number of days on drug (refer section 14.1). A minimum of 80% and a maximum of 120% compliance with the study medication regimen will be required for the patient to considered evaluable per protocol. Subject compliance will be checked through patient diary card and it will be returned to the site at the end of treatment (EOT).

Summary statistics for study medication compliance will be presented by overall and indication using <80%, 80% - 120% and >120% categories with ITT population.

Subject listings of study medication compliance and non-compliance by indication will be presented using ITT population. Each subject will be checked for possible overdosing using the information on maximum recommended dose by body weight provided in APPENDIX 4. Instances of overdosing, if any, will be listed.

## 14.1. DERIVATIONS

Overall percentage of the study intervention compliance will be calculated as follows: Compliance = number of doses taken/ (number of days on therapy x 2) x 100%

## 15. EFFICACY ENDPOINTS

#### 15.1. SECONDARY EFFICACY ENDPOINTS

There are no primary efficacy endpoints defined for this study. The efficacy analysis is defined in terms of secondary and patient diary endpoints.

## Secondary Endpoints -

Early clinical response at the on-therapy visit (Day 3 to 5), defined in terms of 'success'

Document: \\ieedc-vnasc01\BIOSdata\GSK\BRL25000\\PPD\\
Author: \quad \text{Version Number: V1.0} \quad \text{Version Date: \quad 18JUL2022}

Template No.: CS\_TP\_BS016 Revision 6 Reference: CS\_WI\_BS005




- or 'failure' to study intervention.
- Primary clinical response at the end-of-therapy visit (Day 12 to 14), defined in terms of 'success' or 'failure' to study intervention.
- Secondary clinical response at follow-up (Day 22 to 28), defined in terms of 'success' or 'failure' to study intervention.
- Incidence of protocol-defined diarrhea (PDD) in children receiving Augmentin (ES)-600 (AMC/CVA 14:1) at 90/6.4 mg/kg/day in two divided doses administered for 10 days in ARTIs (AOM, ABRS or CABP).

## Definition of clinical responses

Early or Primary Clinical Response will be defined using following criteria: Table 3:

| Success | Clinical cure | Sufficient resolution or improvement of the signs and symptoms such that no additional antibiotic therapy is indicated. |
|---|---|---|
| | Improvement | Improvement in at least 1 presenting sign/symptoms. No additional antibiotic indicated. |
| Failure | Clinical failure | Non-improvement or deterioration in any sign/symptoms after 2 or more days of therapy. Additional antibiotic therapy is indicated. |
| | Unable to determine | A valid assessment of clinical outcome could not be made (eg, participant did not attend or consent to clinical examination or lost to follow-up). |

The proportion of early and primary response will be calculated as follows-

- Proportion of early response = The number of subject who is categorized as success (clinical cure or improvement) at on therapy (OT) visit / the number of subjects in ITT population
- Proportion of primary response = The number of subject who is categorized as success (clinical cure or improvement) at end of therapy (EOT) visit/ the number of subjects in ITT population

Secondary Clinical response will be described using following criteria:

Table 4:

Document: \\ieedc-vnasc01\BIOSdata\GSK\BRL25000\\ \frac{PPD}{PPD} \\ \text{Biostatistics\Documentation\SAP} \\ \text{Version Number: V1.0} \\ \text{Version Date: 18JUL2022} \\ \text{Template No.: CS\_TP\_BS016 Revision 6} \\ \text{Reference: CS\_WI\_BS005} \end{array}

#### Statistical Analysis Plan


| Success | Persistent clinical cure* | Sufficient resolution of signs/symptoms for those Subjects who were clinically cured or improved at the end of therapy. No additional antibiotic indicated. |
|---|---|---|
| Failure | Clinical<br>recurrence | Reappearance of signs/symptoms for those Subjects who were clinically cured or improved at the end of therapy. Additional antibiotic therapy is indicated. |
| | Unable to determine | A valid assessment of clinical outcome could not be made (eg, participant did not attend end of therapy visit, or extenuating circumstances or lost to follow-up). |

<sup>\*</sup> Subjects who showed 'improvement' at EOT (i.e., clinical 'success') and remained same at FU without requiring additional intervention, will be categorized as 'persistent clinical cure'.

The proportion of secondary response will be calculated as follows-

 Proportion of secondary response = The number of subject who is categorized as success (persistent clinical cure) at follow-up (FU) visit / the number of subjects in ITT population

#### Definition of Protocol-defined diarrhoea (PDD)-

The incidence of Protocol-defined diarrhoea (PDD) will be determined based on following rules:

- 3 or more watery stools in one day OR.
- 4 or more loose/watery stools in one day OR
- 2 watery stools per day for two consecutive days OR
- 3 loose/watery stools per day for two consecutive days

#### Patient diary endpoints:

#### Bowel habits

- Mean movement frequency per day
- Maximum movement frequency per day
- Maximum single consistency score

#### Description of Bowel Habits:

Bowel habit ((frequency and consistency of patient's stools) data will be collected using patient diary cards as per schedule of protocol. Bowel movement consistency will be recorded for each patient in five categories —

| Document: | \\ieedc-vnasc01\BIOSdata\GSK\BRL25000\PPD | Biostatistics\Documentation\SAP | | |
|---|---|---|---|---|
| Author: | PPD | | Version Number: | V1.0 |
| TI-4- NI- | . 00 TD D0040 Di-i 0 | | D-f 00 WI D000 | - |

Template No.: CS\_TP\_BS016 Revision 6 Reference: CS\_WI\_BS005



Statistical Analysis Plan




Summary measures of bowel habit movement frequency and consistency are defined as -

- Mean movement frequency per day: this measures the mean number of bowel movements experienced by each patient during the study
- Maximum movement frequency per day: this measures the maximum number of bowel movements experienced in a day for each patient
- Maximum single consistency score: this measures the maximum consistency score for each patient at any time during the study

<u>Clinical Recurrence of Disease</u> - Reappearance of signs/symptoms for those participants who were clinically cured or improved at the end of therapy.

#### 15.1.1. ANALYSIS OF SECONDARY ENDPOINT

## 15.1.1.1. Clinical Response

Frequency and proportion of early, primary, and secondary clinical response will be presented along with 95% CI using exact binomial method

Secondary clinical response statistical analysis will be performed based on as collected data. The following summaries will be generated for early, primary, and secondary clinical response by overall and indication.

- Early clinical response at on-therapy (OT) visit
- Primary clinical response at end of therapy (EOT) visit
- Secondary clinical response at follow-up (FU) visit

Clinical recurrence of disease at follow-up will be summarized with frequency and percentage by overall and indication.

# 15.1.1.2. Incidence of protocol- defined diarrhoea (PDD).

No intercurrent event is defined for this endpoint. The data will be analyzed as collected.

| Document: | \\ieedc-vnasc01\BIOSdata\GSK\BRL25000 PPD | Biostatistics\Documentation\SAP | |
|---|---|---|---|
| Author: | PPD | Version Number: | V1.0 |

Reference: CS\_WI\_BS005

Effective Date: 02Dec2019

Template No.: CS\_TP\_BS016 Revision 6




Frequency and percentage of subjects with incidence of protocol- defined diarrhoea (PDD) will be presented along with 95% CI using exact method (refer SAS code APPENDIX 3)

The following summaries will be generated for incidence of protocol- defined diarrhoea (PDD) by overall and indication.

- Incidence of protocol-defined diarrhoea (PDD)
- Incidence of protocol defined diarrhoea (PDD) over time

Figure for incidence of protocol defined diarrhoea (PDD) over time will also be displayed by overall and indication.

The statistical analysis for incidence of protocol- defined diarrhoea (PDD) will be based on as collected data.

#### 15.1.1.3. Patient diary endpoints

Bowel habits-

The following summaries will be generated for patient summary measures of bowel habit movement by overall and indication.

- Summary and descriptive statistics for patient bowel habit summary measure mean movement frequency per day
- Summary and descriptive statistics for patient bowel habit summary measure maximum movement frequency per day
- Summary and descriptive statistics for patient bowel habit summary measure maximum consistency score

Subject listing of bowel movement by indication will be presented using ITT population.

#### 16. SAFETY ENDPOINTS

All analysis for safety endpoints will be based on the Intent to treat Analysis Set.

#### 16.1. ADVERSE EVENTS

The primary safety endpoint is the number of subjects reporting at least one treatment emergent

Document: \\ieedc-vnasc01\BIOSdata\GSK\BRL25000\\\frac{PPD}{PPD} \\Biostatistics\Documentation\SAP \\
Author: \quad \text{Version Number: V1.0 } \\
Version Date: 18JUL2022 \\
Template No.: CS\_TP\_BS016 Revision 6 \quad \text{Reference: CS\_WI\_BS005}



otatistical Allarysis i la


adverse event (TEAE).

A TEAE duration is defined as an AE which has its onset date during the treatment period + lag time of 1 day.

Adverse Events (AEs) will be coded using MedDRA version 24.1. TEAE's and SAE's will be summarized. All AE's will be listed.

#### 16.1.1. TEAES: PRIMARY SAFETY ENDPOINT

AEs occurring from when a subject sign informed consent to when a subject exits the study will be accounted for in the reporting. AEs occurring pre-treatment, treatment emergent adverse event (on-treatment) and post-treatment periods will be summarized and listed for the ITT population. A treatment -emergent adverse event is defined as any adverse event that develops after initiation of the study treatments or any adverse event already present that worsens following exposure to study treatment.

The primary safety endpoint will be summarized with counts and percentage of subjects reporting any TEAEs and subjects with at least one or any TEAE with corresponding 95% CI using exact binomial method

The following summaries will be generated for adverse events:

- Adverse event overview by period
- Adverse event overview by period for acute otitis media (AOM)
- Adverse event overview by period for acute bacterial rhinosinusitis (ABRS)
- Adverse event overview by period for community acquired bacterial pneumonia (CABP)
- Treatment emergent adverse events by system organ class, preferred term, overall
  and indication
- Adverse events by system organ class, preferred term, overall and indication posttreatment
- Common (>=1%) treatment emergent adverse events by preferred term, overall and indication
- Common (>=1%) adverse events by preferred term, overall and indication posttreatment

AEs and TEAEs will be sorted by descending order of system organ class (SOC) and total frequency of preferred term (PT) within each system organ class (SOC).

Document: \(\left\)\(

Template No.: CS\_TP\_BS016 Revision 6 Reference: CS\_WI\_BS005




AEs and TEAEs related to study drug will presented in decreasing order of preferred term (PT).

Subjects listing of adverse events by indication (TEAE and post-treatment period) will be produced.

#### 16.1.1.1. Severity

Severity is classified as mild, moderate, and severe. An AE with missing severity will be classified as 'Unknown'.

Subjects who experience the same event several times, with different intensities, will only be counted with the maximum intensity.

The following tables will be generated to summarize the severity of adverse event

- Treatment emergent adverse events by system organ class, preferred term, maximum severity, overall and indication
- Adverse events by system organ class, preferred term, maximum severity, overall and indication -post treatment

Sorting order will be presented same as section 16.1.1.

## 16.1.1.2. Relationship to Study Medication

Summary for drug-related treatment emergent adverse events by preferred term, overall and indication will be presented.

# 16.1.2. TEAES LEADING TO PERMANENT DISCONTINUATION OF STUDY MEDICATION OR WITHDRAWAL STUDY

Treatment emergent adverse events leading to permanent discontinuation of study medication or withdrawal from study by system organ class, preferred term, overall and indication will be displayed.

Adverse events leading to withdrawal from study will also be presented by system organ class, preferred term, overall and indication.

Sorting order will be presented same as section 16.1.1.

Subject listing of treatment emergent adverse events leading to permanent discontinuation of study medication or withdrawal from study will also be generated.

Document: \\ieedc-vnasc01\BIOSdata\GSK\BRL25000\\preced{PPD} \Biostatistics\Documentation\SAP \
Author: \quad \text{Version Number: V1.0} \quad \text{Version Date: 18JUL2022}

Template No.: CS\_TP\_BS016 Revision 6 Reference: CS\_WI\_BS005


# 16.1.3. SERIOUS ADVERSE EVENTS

The following summaries will be presented for serious adverse events:

- Treatment emergent serious adverse events by system organ class, preferred term, overall
  and indication
- Serious adverse events by system organ class, preferred term, overall and indication post-treatment
- Treatment emergent serious adverse events by system organ class and preferred term, maximum severity, overall and indication
- Serious adverse events by system organ class, preferred term, maximum severity, overall and indication -post treatment
- Drug-related treatment emergent serious adverse events by preferred term, overall and indication

Sorting order will be presented same as section 16.1.1.

The following serious adverse event listings will be produced:

- Listing of reasons for considering as a serious adverse event by indication- pre-treatment
- Listing of fatal and non-fatal serious adverse events (TEAE and post-treatment period)
- Listing of reasons for considering as a serious adverse event by indication (TEAE and post-treatment period)

#### 16.1.4. ADVERSE EVENTS LEADING TO DEATH

Subject listing will be generated for adverse event leading to death.

#### 16.1.5. . CARDIOVASCULAR EVENTS

The following AE's/SAE's will be classified as Cardiovascular events:

- Myocardial infarction/unstable angina
- Congestive heart failure
- Arrhythmias
- Valvulopathy
- Pulmonary hypertension

Document: \\ieedc-vnasc01\BIOSdata\GSK\BRL25000\\frac{PPD}{Version Number: V1.0}
\text{Version Date: 18JUL2022}

Template No.: CS\_TP\_BS016 Revision 6 Reference: CS\_WI\_BS005




- Cerebrovascular events/stroke and transient ischemic attack
- Peripheral arterial thromboembolism
- Deep venous thrombosis/pulmonary embolism
- Revascularization

Subject listing will be generated for all cardiovascular events recorded in the study.

### **16.2. DEATHS**

Subject listing will be generated for any death that happens during the study.

### 16.3. LABORATORY EVALUATIONS

Laboratory parameters assessed for the study are listed below:

#### Table 5:

| Assessments | Parameters | | |
|---|---|---|---|
| Hematology | Platelet Count RBC Count Hemoglobin Hematocrit | RBC Indices:<br>MCV<br>MCH<br>%Reticulocytes | WBC count with Differential: Neutrophils Lymphocytes Monocytes Eosinophils Basophils |
| Clinical<br>Chemistry | Plasma<br>creatinine | Aspartate<br>Aminotransferase (AST)<br>Alanine<br>Aminotransferase<br>(ALT) | Total and direct<br>bilirubin |
| Radiography | Chest X ray to be performed for patients presumed to a diagnosis of CABP. X ray of nasal/paranasal sinus to be performed for patients presumed to have ABRS (both only for reference, as per investigators discretion) | | |

 Clinical laboratory evaluations include hematology, clinical chemistry, A list of laboratory assessments is mentioned in Table 5which will be used for statistical analysis.

Descriptive statistics (n, mean, standard deviation (SD), median, minimum value

Document: \\ieedc-vnasc01\BIOSdata\GSK\BRL25000\\preced{PPD} Biostatistics\Documentation\SAP


Template No.: CS\_TP\_BS016 Revision 6 Reference: CS\_WI\_BS005




(min), and maximum value (max)) will be presented for quantitative measurements of laboratory parameters by overall and indication, Frequency and percentage will be displayed for qualitative measurements of laboratory parameters by overall and indication.

Subjects listing of baseline laboratory parameters by indication will also be generated.

### 16.4. ECG EVALUATIONS

ECG assessment will not be performed for this study.

### 16.5. VITAL SIGNS

The following Vital Signs measurements will be reported for this study:

- Respiratory Rate (breaths/min)
- Temperature (° C)
- Pulse rate
- Weight (kg)
- Height

Actual vital signs results, change from baseline values and percentage change from baseline will be summarized for each analysis visit.

Subjects listing of vital signs parameters by indication will also be generated.

### 16.6. OTHER SAFETY ASSESSMENTS

Summary for visits impacted by COVID-19 pandemic will be presented by overall and indication.

Subject listing of Covid-19 pandemic study impact (TEAE and post-treatment period) will be displayed.

Subject listing of local examination by indication will be generated.

\\ieedc-vnasc01\BIOSdata\GSK\BRL25000\PPD Biostatistics\Documentation\SAP Document: PPD Author: Version Number: V1.0 Version Date: 18JUL2022

Template No.: CS\_TP\_BS016 Revision 6 Reference: CS\_WI\_BS005



Statistical Analysis Plan 

Subject listing will be generated for pregnancy.

#### DATA NOT SUMMARIZED OR PRESENTED **17.**

Not applicable

#### **18**. REFERENCES

Protocol number 213514 | Protocol Amendment 01 19 May 2021.

\\ieedc-vnasc01\BIOSdata\GSK\BRL25000\PPD Biostatistics\Documentation\SAP Document: PPD

Author: Version Number: V1.0 Version Date: 18JUL2022

Reference: CS\_WI\_BS005

Template No.: CS\_TP\_BS016 Revision 6




213514

### APPENDIX 1. Programming Conventions for Outputs

### IQVIA OUTPUT CONVENTIONS

Outputs will be presented according to IQVIA Global Biostatistics Standard Output Conventions

#### DATES & TIMES

Depending on data available, dates and times will take the format DDMMMYYYY; times will format HH.MM combined dates and times will take the format DDMMMYYYY/HH:MM. Time will be based on a 24 hour clock.

### SPELLING FORMAT

English UK, including for MedDRA where British English is used.

#### LISTINGS

All listings will be ordered by the following (unless otherwise indicated in the template):

- Subject ID
- Date and time (where applicable)

#### PRESENTATION OF TREATMENT GROUPS

For outputs, treatment groups will be represented as follows:

Treatment Group Augmentin (ES) – 600

### DESCRIPTIVE STATISTICS

If the original data has N decimal places, then the summary statistics will have the following decimal places:

\\ieedc-vnasc01\BIOSdata\GSK\BRL25000 PPD Biostatistics\Documentation\SAP Document: Author: Version Number: V1.0 Version Date: 18JUL2022

Template No.: CS\_TP\_BS016 Revision 6 Reference: CS\_WI\_BS005



Statistical Analysis Plan


- Minimum and maximum: N;
- Mean, median, lower and upper bounds of two-sided 95% CI: N + 1;
- SD and SE: N + 2

#### PERCENTAGES

Percentages will be reported to one decimal place. Rounding will be applied, except for percentages < 0.1 but > 0.0 which will be presented as '< 0.1' and percentages < 100.0 but >99.9 which will be presented as '>99.9'.

Where counts are zero, no percentages will appear in the output.

Document: \\ieedc-vnasc01\BIOSdata\GSK\BRL25000\\protector\PD \\Biostatistics\Documentation\SAP


Template No.: CS\_TP\_BS016 Revision 6 Reference: CS\_WI\_BS005




### APPENDIX 2. Partial Date Conventions

Date Imputation Rule for adverse events and concomitant medication for assigning the event in particular period:

Missing day in a start date, e.g. - -JUN2021, set to the first of the month, 01JUN2021.

Missing month in a start date, e.g., 15- - -2006, set to January, 15JAN2021.

Missing day in a stop date, e.g. - -APR2021, set to the last of the month, 30APR2021.

Missing month in a stop date, e.g., 23- - -2006, set to December, 23DEC2021.

If both day and month are missing, e.g. - - - - -2021, apply both rules giving 01JAN2021 for a partial start date, or 31DEC2021 for a partial stop date

Document: \\ieedc-vnasc01\BIOSdata\GSK\BRL25000\\PPD \\Biostatistics\Documentation\SAP


Template No.: CS\_TP\_BS016 Revision 6 Reference: CS\_WI\_BS005

Complate No.: 00\_11 \_D0010 Nevision 0




## APPENDIX 3. SAS CODE FOR ANALYSES

The following SAS code will be used to analyze the clinical response:

### For overall:

```
proc freq data=modeldata;
tables response/binomial (exact) alpha=0.05;
output out= ci95 binomial
run;
```

### For indication wise analysis

```
proc freq data=modeldata;
by indication
tables response/binomial (exact) alpha=0.05;
output out= ci95 binomial
run:
```

Note: In the absence of responder category (zero responder), separate category with zero responder in final data set will be added before passing in proc freq using Weight statement with zeroes option as below

SAS code: proc freq data=modeldata; by indication; tables response / binomial; weight wgt/zeroes; exact binomial; run:

\\ieedc-vnasc01\BIOSdata\GSK\BRL25000\PPD Biostatistics\Documentation\SAP Document: Author: Version Number: V1.0

Version Date:

18JUL2022

Template No.: CS\_TP\_BS016 Revision 6 Reference: CS\_WI\_BS005




# APPENDIX 4. MAXIMUM RECOMMENDED DOSE BY BODY WEIGHT

| Body weight (kg) # | Augmentin 600<br>for oral<br>suspension (ml)<br>twice in<br>day(BID) | Maximum Recommended Dose Administered by the Oral Route (ml) Twice in day(BID) | | Augmentin 600<br>for oral<br>suspension (ml)<br>twice in<br>day(BID) | Maximum Recommended Administered by the Oral Route (ml) Twice in day(BID) |
|---|---|---|---|---|---|
| | | | 21 | 8.0 | 10.5 |
| | | | 22 | 8.4 | 11.0 |
| 3 | 1.2 | 1.5 | 23 | 8.6 | 11.5 |
| 4 | 1.6 | 2.0 | 24 | 9.0 | 12.0 |
| 5 | 2.0 | 2.5 | 25 | 9.4 | 12.5 |
| 6 | 2.4 | 3.0 | 26 | 9.8 | 13.0 |
| 7 | 2.6 | 3.5 | 27 | 10.2 | 13.5 |
| 8 | 3.0 | 4.0 | 28 | 10.6 | 14.0 |
| 9 | 3.4 | 4.5 | 29 | 11.0 | 14.5 |
| 10 | 3.8 | 5.0 | 30 | 11.4 | 15.0 |
| 11 | 4.2 | 5.5 | 31 | 11.6 | 15.5 |
| 12 | 4.6 | 6.0 | 32 | 12.0 | 16.0 |
| 13 | 5.0 | 6.5 | 33 | 12.4 | 16.5 |
| 14 | 5.4 | 7.0 | 34 | 12.8 | 17.0 |
| 15 | 5.6 | 7.5 | 35 | 13.2 | 17.5 |
| 16 | 6.0 | 8.0 | 36 | 13.6 | 18.0 |
| 17 | 6.4 | 8.5 | 37 | 14.0 | 18.5 |
| 18 | 6.8 | 9.0 | 38 | 14.4 | 19.0 |
| 19 | 7.2 | 9.5 | 39 | 14.6 | 19.5 |
| 20 | 7.6 | 10.0 | 40 | 15.0 | 20.0 |

Document: \\ieedc-vnasc01\BIOSdata\GSK\BRL25000 PPD \\Biostatistics\Documentation\SAP


Template No.: CS\_TP\_BS016 Revision 6 Reference: CS\_WI\_BS005

Effective Date: 02Dec2019

Copyright © 2009, 2010, 2012, 2016, 2018, 2019 IQVIA. All rights reserved. The contents of this document are confidential and proprietary to IQVIA Holdings Inc. and its subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.

| | | | D | ocuSign |
|---|---|---|---|---|
| Certificate Of Completion | | | | |
| Envelope Id: PPD | | | Status: Completed | |
| Subject: Please DocuSign: GSK_213514 SAP | | | | |
| Project Code (Enter 0 for non-billable projects) IQVIA ID (Login ID): | ): | | | |
| Business Unit: | | | | |
| DSSR | | | | |
| Source Envelope: | | | | |
| Document Pages: 43 | Signatures: 5 | | Envelope Originator: | _ |
| Certificate Pages: 6 | Initials: 0 | Pi | PD | |
| AutoNav: Enabled | | | | |
| Envelopeld Stamping: Disabled Time Zone: (UTC-05:00) Eastern Time (US & | Canada) | | | |
| Time Zone. (010-03.00) Lasterii Time (03 d | Canada) | | | |
| B | DDD | | | |
| | PPD | | | |
| Status: Original<br>7/18/2022 5:40:27 AM | | | Location: DocuSign | |
| 7710/2022 3.40.27 AWI | | | | |
| Signer Events | Signature | | Timestamp | |
| | | | Sent: 7/18/2022 5:47:45 AM | |
| | | | Viewed: 7/18/2022 6:02:33 AM | |
| | | | Signed: 7/18/2022 6:03:18 AM | |
| | W. C | . 5 6: | | |
| | With Signing Authenticatio<br>With Signing Reasons (on | | word | |
| | I am the author of this do | • | | |
| Electronic Record and Signature Disclosure | | | | |
| Accepted: 7/18/2022 6:04:10 AM<br>PPD | | | | |
| Company Name: IQVIA | | | | |
| D | PPD | | C | |
| | | | Sent: 7/18/2022 5:47:47 AM<br>Viewed: 7/18/2022 5:53:41 AM | |
| IQVIA Biotech DocuSign Part 11 | | | Signed: 7/18/2022 5:54:05 AM | |
| Security Level: Email, Account Authentication | | | | |
| (Required), Logged in | Signature Adoption: Pre-se<br>PPD | elected Style | _ | |
| | | | _ | |
| | With Signing Authentication | | eword | |
| | With Signing Reasons (on | | | |
| | I am the author of this do | ocument | | |

Electronic Record and Signature Disclosure: Not Offered via DocuSign

Signer Events Signature PPD

Sent: 7/18/2022 5:47:47 AM Viewed: 7/18/2022 8:45:24 AM Signed: 7/18/2022 8:49:29 AM

Timestamp

With Signing Authentication via DocuSign password With Signing Reasons (on each tab): I approve this document

Electronic Record and Signature Disclosure: Accented: 7/18/2022 8:45:24 AM
PPD

Company Name: IQVIA

PPD

PPD

Sent: 7/18/2022 5:47:49 AM Viewed: 7/18/2022 6:28:02 AM Signed: 7/18/2022 6:29:33 AM

With Signing Authentication via DocuSign password With Signing Reasons (on each tab): I am the author of this document

Electronic Record and Signature Disclosure:

Accepted: 7/18/2022 6:28:02 AM PPD

Company Name: IQVIA

Sent: 7/18/2022 5:47:49 AM

Viewed: 7/20/2022 6:15:25 AM Signed: 7/20/2022 6:16:47 AM

With Signing Authentication via DocuSign password With Signing Reasons (on each tab): I approve this document

Electronic Record and Signature Disclosure:

Accepted: 7/20/2022 6:15:25 AM PPD

Company Name: IQVIA

In Person Signer Events Signature Timestamp **Editor Delivery Events** Status Timestamp Timestamp Agent Delivery Events Status Intermediary Delivery Events Status Timestamp **Certified Delivery Events Status** Timestamp

| Carbon Copy Events | Status | Timestamp |
|---|---|---|
| Witness Events | Signature | Timestamp |
| Notary Events | Signature | Timestamp |
| Envelope Summary Events | Status | Timestamps |
| Envelope Sent | Hashed/Encrypted | 7/18/2022 5:47:49 AM |
| Certified Delivered | Security Checked | 7/20/2022 6:15:25 AM |
| Signing Complete | Security Checked | 7/20/2022 6:16:47 AM |
| Completed | Security Checked | 7/20/2022 6:16:47 AM |
| Payment Events | Status | Timestamps |
| Electronic Record and Signature Disclosure | | |

### CONSENT TO ELECTRONIC DELIVERY AND EXECUTION OF DOCUMENTS

From time to time, IQVIA ("we" or "us") may provide you certain written contracts, notices, disclosures, authorizations, acknowledgements or other documents (collectively, the "Documents") electronically. Please read this consent form carefully. It explains the terms and conditions under which such Documents are provided by us and executed by you electronically through your DocuSign, Inc. ("DocuSign") user account. If you consent to the delivery and execution of such Documents electronically, please click the "I Agree" button.

### **Documents will be sent to you electronically**

If you consent to electronic delivery, Documents will be sent to your DocuSign user account. You may request a paper copy of documents previously made available through your DocuSign user account, but an additional charge may be incurred. Alternatively, you can download and print documents sent to your DocuSign user account. Unless otherwise noted, you can access a Document up to 30 days from the date we first sent the Document to you.

### Withhold Consent or Withdrawing Consent to Electronic Delivery

If you withhold consent to electronic delivery or execution, or withdraw your consent at a later date, all Documents will be sent to your mailing address following our receipt of notice of such action. The following sections explain the consequences of withholding or withdrawing your consent to electronic delivery and execution of Documents, and also the procedures you must follow in order to effectuate delivery to your mailing address.

### **Consequences of Withdrawing Consent**

By electing to only receive and execute Documents sent to your mailing address, we will not be able to carry out transactions or services as efficiently. For instance, some transactions or services require your express consent. We can perform these transaction or services only if we first receive an acknowledgement that indicates you received and consent to the Document related to the proposed transaction or service.

To withhold consent now or withdraw consent at a later date, please sign DocuSign's "Withdraw Consent" form on the signing page of your DocuSign user account. This will indicate that you have withdrawn your consent to receive Documents electronically. Once you sign the "Withdraw Consent" form, you will no longer be able to use your DocuSign user account to execute Documents electronically and we will send Documents to your mailing address. Withdrawal of consent does not affect the validity of any Documents previously executed electronically prior to such withdrawal of Consent. In addition, should you execute any Documents electronically, your execution of such Documents shall indicate your continued consent to execute such Documents electronically.

#### **How to contact IOVIA:**

If you would like us to send the Documents to a different e-mail address, request paper copies of Documents you have previously received electronically, or withdraw your consent to receive electronic documents, please follow the instructions below. If you have any other questions, please contact: DocuSignSupport@IQVIA.com

### 1. To advise IQVIA of your new e-mail address

If you would like your Documents sent to a different e-mail address, you must send an e-mail message to DocuSignSupport@IQVIA.com . In the body of the e-mail please state the following: (i) your previous e-mail address, and (ii) your new e-mail address. No other information is required.

In addition, you must notify DocuSign of your new e-mail address. Please log into your DocuSign user account, and follow the instructions to update your e-mail address.

### 2. To request paper copies from IQVIA

To request paper copies of Documents you have received previously through your DocuSign user account, send an e-mail to DocuSignSupport@IQVIA.com

In the body of the e-mail please state the following: (i) your e-mail address, (ii) full name, (iii) U.S. Postal address, and (iv) telephone number. Additional charges may apply for such paper copies.

### 3. To withdraw your consent with IQVIA

To withdraw your consent to receiving and executing Documents in an electronic format, you may do one of the following:

i. decline to sign a document from within your DocuSign user account, and on the subsequent page, select the check-box indicating you wish to withdraw your consent; or ii. send us an e-mail to DocuSignSupport@IQVIA.com and in the body of such request you must state your e-mail, full name, US Postal Address, telephone number, and account number. No additional information is necessary.

### Required hardware and software

| Operating Systems: | Windows® 2000, Windows® XP, Windows Vista®; Mac OS® X |
|---|---|
| Browsers: | <ul> <li>Internet Explorer (Windows Only) 8.0 or above – compatibility mode is supported only for 9.0 and above.</li> <li>Windows Edge Current Version</li> <li>Mozilla Firefox Current Version</li> <li>Safari (Mac OS only) 6.2 or above</li> <li>Google Chrome Current Version</li> </ul> |
| PDF Reader: | Acrobat® or similar software may be required to view and print PDF files |
| Screen Resolution: | 1024 x 768 Recommended |
| Enabled Security Settings: | Allow per session cookies |
| Mobile Signing: | <ul><li>Apple iOS 7.0 or above</li><li>Android 4.0 or above</li></ul> |

<sup>\*\*</sup> These minimum requirements are subject to change. If these requirements change, we will provide you with an e-mail message at the e-mail address we have on file for you at the time the hardware and software requirements are revised.

Pre-release (e.g. beta) versions of operating systems and browsers are not supported.

### Acknowledging your access and consent to receive materials electronically

To confirm you can access this information electronically and that you consent to receiving and executing Documents electronically on the terms and conditions described above, please let us know by clicking the "I Agree" button.

By clicking the "I Agree" button, you confirm that

- You can access and read this Consent To Electronic Delivery and Execution of Documents; and
- You can print on paper the disclosure or save or send the disclosure to a place where you can print it, for future reference and access; and
- Until or unless you notify IQVIA as described above, you consent to the delivery and execution of Documents electronically.

# Signature Page for $\,213514$ TMF-14854664 $\,v1.0$

| | PPD |
|---|---|
| Reason for signing: Approved | Name: |
| | Role: Approver |
| | Date of signature: 21-Jul-2022 10:35:21 GMT+0000 |

Signature Page for TMF-14854664 v1.0